CLINICAL TRIAL: NCT02016703
Title: Gastrointestinal Tolerance of Erythritol-containing Beverages in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CER-TDEOH05
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2013-12

CONDITIONS: Gastrointestinal; Tolerance
Keywords: erythritol; polyol; laxation; gastrointestinal; tolerance; soft drinks; child; diarrhoea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 5 g group (Experimental): 5g erythritol dissolved in 250 ml (2% w/v) consumed within 15 min between meals (tested vs. 250 ml isosweet saccharose placebo under same conditions)
  Interventions: Other: Erythritol drink; Other: Placebo drink
- 15 g group (Experimental): 15g erythritol dissolved in 250 ml (6% w/v) consumed within 15 min between meals (tested vs. 250 ml isosweet saccharose placebo under same conditions)
  Interventions: Other: Erythritol drink; Other: Placebo drink
- 25 g group (Experimental): 25g erythritol dissolved in 250 ml (10% w/v) consumed within 15 min between meals (tested vs. 250 ml isosweet saccharose placebo under same conditions)
  Interventions: Other: Erythritol drink; Other: Placebo drink
- 20 g group (Experimental): 20g erythritol dissolved in 250 ml (8% w/v) consumed within 15 min between meals (tested vs. 250 ml isosweet saccharose placebo under same conditions)
  Interventions: Other: Erythritol drink; Other: Placebo drink

INTERVENTIONS:
Other: Erythritol drink
Other: Placebo drink

SUMMARY:
Purpose of this study: assess the maximum tolerated bolus dose of erythritol, delivered in a clear beverage, compared with placebo (saccharose) in 4-6 year old children.

DETAILED DESCRIPTION:
The study is a randomized placebo-controlled, double-blind cross-over trial designed to determine the gastrointestinal (GI) responses and maximum tolerated dose of erythritol in young children as a single oral dose in a beverage in-between meals.

The children were divided into 4 dose groups. In each group of children, only one dose level was tested such that each child was exposed to only a single dose level versus placebo. The erythritol dose started at 5 grams and was increased by 10 g between each group of children only if the preceding dose level was found to have no significant GI tolerance effects. The effects on faecal parameters and gastrointestinal complaints were recorded in order to determine the threshold dose. After finding a significant difference in tolerance between erythritol and placebo in the 25 g dose cohort, a protocol amendment was approved allowing the investigators to study a dose of 20 g.

Test materials were prepared by Cargill, Vilvoorde, Belgium and supplied in bottles containing 250 mL of a noncarbonated fruit-flavoured (two flavours: strawberry and orange) clear drink sweetened with erythritol at four different dose levels: 5, 15, 20 and 25 g (equivalent to 2, 6, 8 and 10% w/v erythritol, respectively). Placebo was supplied in an identical manner but prepared with common nutritive carbohydrates (saccharose and maltodextrin) and providing an equivalent sweetness to that of the corresponding erythritol beverages (i.e.: 1.4, 4.2, 5.6 and 7% w/v).

In total 185 healthy young children aged 4-6 years were recruited at three clinical investigation centres after informed consent of both parents; 184 completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 4 to 6 years at Study D1 (day of consumption of the first beverage)
* Body Mass Index ³ 13 kg/m²
* Accustomed to having breakfast
* Having a regular defecation frequency inferior or equal to two per day
* Able to drink 250 mL within 15 minutes
* Toilet-trained / able to use a potty (both at day and night)
* Informed consent of both person entitled to parental rights
* Person entitled to parental rights affiliated to the French social security

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before D1 of the study
* Participation in any non-invasive clinical trial up to 30 days before D1 of this study, including blood sampling and/ or, intravenous, inhalatory administration of substances
* Having a history of medical or surgical events that may significantly affect the study outcome, such as gastric and digestive diseases
* Any current metabolic or endocrine disease, including diabetes mellitus
* Use of medication, including antibiotics, laxatives and steroids
* Regular gastrointestinal complaints, such as stomach upsets, diarrhoea, constipation, flatulence, abdominal colic

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Diarrhoea and/or significant gastrointestinal (GI) symptoms | 48 hours
  Diarrhoea = a single watery stool (Bristol Stool Scale Score of 7) and/or >3 faeces (regardless of consistency) in a 24 h period.
  Significant GI symptoms = any GI symptoms having a severity recorded as "severe intensity" in the symptom diary

SECONDARY OUTCOMES:
Stool frequency | 48 hours
Stool consistency | 48 hours
  Stools were assigned a consistency score using the Bristol Stool Scale
Gastrointestinal symptoms | 24 hours
  Occurrence, intensity and frequency of borborygmi, excess flatus, abdominal pain, distended stomach (bloating) and nausea. For vomiting, information collected included occurrence and frequency. Symptom intensity was graded as 0 (none), 1 (mild), 2 (average) and 3 (severe) except for vomiting.
Urinary erythritol excretion | 24 hours
  Urine was collected for 24 h after consumption of the test drink and analyzed by HPLC to estimate the proportion absorbed and excreted.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Jacqz-Aigrain, PhD, Principal Investigator — Clinical Investigation Centre Robert Debré Hospital, Paris, France
Locations (3):
- France (3):
  - Clinical Investigation Centre Louis Pradel Hospital, Bron
  - Biofortis Merieux NutriSciences, Nantes
  - Clinical Investigation Centre Robert Debré Hospital, Paris

REFERENCES:
- [Background] Bornet FR, Blayo A, Dauchy F, Slama G. Plasma and urine kinetics of erythritol after oral ingestion by healthy humans. Regul Toxicol Pharmacol. 1996 Oct;24(2 Pt 2):S280-5. doi: 10.1006/rtph.1996.0109. PMID 8933644
- [Background] Arrigoni E, Brouns F, Amado R. Human gut microbiota does not ferment erythritol. Br J Nutr. 2005 Nov;94(5):643-6. doi: 10.1079/bjn20051546. PMID 16277764
- [Background] Bornet FR, Blayo A, Dauchy F, Slama G. Gastrointestinal response and plasma and urine determinations in human subjects given erythritol. Regul Toxicol Pharmacol. 1996 Oct;24(2 Pt 2):S296-302. doi: 10.1006/rtph.1996.0111. PMID 8933646
- [Background] Tetzloff W, Dauchy F, Medimagh S, Carr D, Bar A. Tolerance to subchronic, high-dose ingestion of erythritol in human volunteers. Regul Toxicol Pharmacol. 1996 Oct;24(2 Pt 2):S286-95. doi: 10.1006/rtph.1996.0110. PMID 8933645
- [Background] Munro IC, Berndt WO, Borzelleca JF, Flamm G, Lynch BS, Kennepohl E, Bar EA, Modderman J. Erythritol: an interpretive summary of biochemical, metabolic, toxicological and clinical data. Food Chem Toxicol. 1998 Dec;36(12):1139-74. doi: 10.1016/s0278-6915(98)00091-x. PMID 9862657
- [Background] Storey D, Lee A, Bornet F, Brouns F. Gastrointestinal tolerance of erythritol and xylitol ingested in a liquid. Eur J Clin Nutr. 2007 Mar;61(3):349-54. doi: 10.1038/sj.ejcn.1602532. Epub 2006 Sep 20. PMID 16988647
- [Background] Lifshitz F, Ament ME, Kleinman RE, Klish W, Lebenthal E, Perman J, Udall JN Jr. Role of juice carbohydrate malabsorption in chronic nonspecific diarrhea in children. J Pediatr. 1992 May;120(5):825-9. doi: 10.1016/s0022-3476(05)80260-4. No abstract available. PMID 1578324
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672